CLINICAL TRIAL: NCT01045954
Title: A Study of the Rules for Insulin Dosing in Patients Using Multiple Daily Injections
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Diabetes Care Center (Industry)
Responsible Party: Allen B. King, MD, Diabetes Care Center
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: DCC 02-09
Record Dates: First submitted 2010-01-07; First posted 2010-01-11 (Estimated); Last update posted 2010-01-11 (Estimated); Status verified 2010-01

CONDITIONS: Diabetes Mellitus Type 1
Keywords: diabetes mellitus type 1; continuous glucose monitoring
MeSH Terms: conditions — Diabetes Mellitus, Type 1 | interventions — Insulin Lispro; Insulin Glargine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Lispro Insulin and glargine insulin — Continuous glucose sensor will be inserted. Subject will be on an isocaloric diet and CGM downloaded daily. Insulin basal and bolus will be adjusted based upon treatment goals until goals reached

SUMMARY:
This study will be conducted in subjects with Type 1 diabetes mellitus on multiple daily insulin injections to determine the correct insulin dosing formulas. Subjects will be evaluated using continuous glucose monitoring.

DETAILED DESCRIPTION:
Subjects with stable type 1 diabetes mellitus on multiple daily insulin injections including basal and bolus will be selected in order to determine the correct insulin dosing formulas. Subjects will be placed on continuous glucose sensor (CGMS) and an isocaloric diet. Subjects will have the CGMS downloaded daily and the insulin doses adjusted if necessary. Subject will do four SMBGs daily to calibrate CGMS and on last day a 7-point SMBG. subjects will be on lispro and glargine insulin. Basal insulin will be once a day.

ELIGIBILITY:
Inclusion Criteria:

* Age: >17 years
* Type 1 diabetes
* Diabetes duration > 3 months
* On treatment with multiple daily injections either one or more basal insulin injections each day for 6 weeks
* HbA1c <9.0%
* Stable HbA1c in the proceeding 3 months (i.e., change <1%)
* Demonstrated adherence to visits and instructions
* Attend a class in meal carbohydrate content estimation or have demonstrated knowledge of carbohydrate counting

Exclusion Criteria:

* Major stress event during or for 6 weeks before the evaluation
* Taking a medication that can alter insulin sensitivity
* Within one week of menses
* Unstable eating or activity pattern
* Pregnancy
* Weight gain of > 1.5 kg during the preceding 3 months
* Serum creatinine of >1.5 mg/dl
* Active liver disease
* Evidence of autonomic neuropathy, especially gastroparesis
* Any antidiabetic medication other than insulin
* Treatment with continuous subcutaneous insulin infusion

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2010-01; Primary Completion 2010-08 (Estimated); Study Completion 2010-10 (Estimated)

PRIMARY OUTCOMES:
Determine the mean value for the slop between the variables of total daily dose versus total basal dose. | Two weeks

SECONDARY OUTCOMES:
Determine the slope between the other variables: weight, total daily dose, total basal dose, insulin correction carbohydrate rate, correction factor | Two weeks

CONTACTS AND LOCATIONS:
Overall Officials: Allen B. King, MD, Principal Investigator — Diabetes Care Center
Locations (1):
- Diabetes Care Center, Salinas, California, United States

REFERENCES:
- [Background] Walsh J, Roberts R. Pumping Insulin. 3rd Edition, San Diego, Torrey Pines Press. 2000
- [Background] Bode BW. Insulin Pump Therapy. In, Therapy for diabetes Mellitus and Related Disorders, fourth edition, Lebovitz H. Ed, Alexandria, VA, American Diabetes Association, 2004, p224-231
- [Background] King AB, Armstrong DU. A prospective evaluation of insulin dosing recommendations in patients with type 1 diabetes at near normal glucose control: bolus dosing. J Diabetes Sci Technol. 2007 Jan;1(1):42-6. doi: 10.1177/193229680700100107. PMID 19888378
- [Background] King AB, Armstrong DU. A prospective evaluation of insulin dosing recommendations in patients with type 1 diabetes at near normal glucose control: Basal dosing. J Diabetes Sci Technol. 2007 Jan;1(1):36-41. doi: 10.1177/193229680700100106. PMID 19888377
- [Background] Davidson PC, Hebblewhite HR, Bode BW, et al. Statistically based CSII parameters correction factor, CF (1700 rule) carbohydrate-to-insulin ratio, CIR (2.8 rule) and basal-to-total ration. Diabetes Technol Ther. 2003; 3:237